CLINICAL TRIAL: NCT01984372
Title: A Multi-centre, Open Label, Observational, Non-interventional, Post Marketing Surveillance to Evaluate Safety and Effectiveness During Long-term Treatment With Tresiba® (Insulin Degludec) in Patients With Diabetes Mellitus Requiring Insulin Therapy Under Normal Clinical Practice Conditions
Brief Title: Post-marketing Surveillance (Special Use-results Surveillance) on Long-term Use With Tresiba®
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN1250-4061; U1111-1144-4412 (Other: WHO)
Record Dates: First submitted 2013-11-07; First posted 2013-11-14 (Estimated); Last update posted 2020-08-04 (Actual); Status verified 2020-08

CONDITIONS: Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — insulin degludec

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Tresiba® users
  Interventions: Drug: insulin degludec

INTERVENTIONS:
Drug: insulin degludec — Frequency and timing of visits are based on normal clinical practice for patients with diabetes mellitus requiring insulin therapy.

SUMMARY:
This study is conducted in Asia. The aim of this post marketing surveillance (PMS) is to assess safety and effectiveness of long-term treatment with Tresiba® (insulin degludec) in patients with diabetes mellitus requiring insulin therapy under normal clinical practice conditions.

A total of 4000 patients will be enrolled to investigate long term (3 years of treatment) safety of Tresiba® and additional 2000 patients will be enrolled to assess the safety in an early stage of the PMS more precisely. At the time of enrolment the patients will be randomly allocated to either 3 years or 6 months observation group.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diabetes mellitus requiring insulin therapy for whom the treating physician has decided to start Tresiba® treatment

Exclusion Criteria:

* Patients who are or have previously been on Tresiba® therapy
* Patients who have previously been participating in this PMS

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with diabetes mellitus requiring insulin therapy not previously treated with Tresiba®, including newly-diagnosed patients whom the physician has judged as appropriate to start treatment with Tresiba®.
Sampling Method: Non-Probability Sample
Enrollment: 6163 (Actual)
Dates: Start 2013-11-06 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Incidence of AEs (Adverse Events) by preferred term | During 3 years of treatment

SECONDARY OUTCOMES:
Incidence of AEs (Adverse Events) by preferred term | During 6 months of treatment
Incidence of SADRs (Serious Adverse Drug Reactions) by preferred term | During 6 months of treatment
Incidence of SADRs (Serious Adverse Drug Reactions) by preferred term | During 3 years of treatment
Incidence of serious allergic reactions (systemic or localized, including injection site reactions) by preferred term | During 6 months of treatment
Incidence of serious allergic reactions (systemic or localized, including injection site reactions) by preferred term | During 3 years of treatment
Incidence of severe hypoglycaemia | During 6 months of treatment
Incidence of severe hypoglycaemia | During 3 years of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Tokyo, Japan

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com